CLINICAL TRIAL: NCT03016949
Title: A Phase 3, Open-label, Randomized Trial to Evaluate Humoral Immunogenicity of Various Schedules of Intramuscular Full Dose and Intradermal Fractional Dose of Inactivated Polio Vaccine in Infants
Brief Title: A Study to Evaluate Immunogenicity of Various Schedules of Inactivated Polio Vaccine
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Regulatory timelines for approval expired
Sponsor: Fidec Corporation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IPV-003-ABMG
Record Dates: First submitted 2017-01-05; First posted 2017-01-11 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A (Experimental): 3 doses IPV IM at 10, 14 & 36 weeks of age incl. blood sampling at 10, 18, 36 & 40 weeks.
  Interventions: Biological: IPV
- Group B (Experimental): 3 doses f-IPV ID at 10, 14 & 36 weeks of age incl. blood sampling at 10, 18, 36 & 40 weeks.
  Interventions: Biological: f-IPV
- Group C (Experimental): 2 doses IPV IM at 14 & 36 weeks of age incl. blood sampling at 14, 18, 36 & 40 weeks.
  Interventions: Biological: IPV
- Group D (Experimental): 2 doses f-IPV ID at 14 & 36 weeks of age incl. blood sampling at 14, 18, 36 & 40 weeks.
  Interventions: Biological: f-IPV
- Group E (Experimental): 3 doses IPV IM at 6, 14 & 36 weeks of age incl. blood sampling at 6, 18, 36 & 40 weeks.
  Interventions: Biological: IPV
- Group F (Experimental): 3 doses f-IPV ID at 6, 14 & 36 weeks of age incl. blood sampling at 6, 18, 36 & 40 weeks.
  Interventions: Biological: f-IPV

INTERVENTIONS:
Biological: IPV — Comparison of different vaccination schedules with 2 different vaccines (IPV and f-IPV) and 2 different types of administration (IM and ID)
  Arms: Group A; Group C; Group E
Biological: f-IPV — Comparison of different vaccination schedules with 2 different vaccines (IPV and f-IPV) and 2 different types of administration (IM and ID)
  Arms: Group B; Group D; Group F

SUMMARY:
The study will evaluate the humoral immunogenicity in various schedule combinations of full dose inactivated polio vaccines (IPV) via intramuscular administration (IM) and of the fractional dose of inactivated poliovaccine (f-IPV) via intradermal administration (ID).

DETAILED DESCRIPTION:
The study will be conducted in a setting where only IPV is being used for polio prevention in infant immunization schedules.

The study population will include infants from Uruguay, a pioneer country in immunization programs in Latin America, where tOPV(trivalent oral polio vaccine) was used until 2012, after which the program changed to an all-IPV schedule without transition.

The primary IPV immunization schedule in the country is as stand-alone vaccine at 2, 4 and 6 months of age, with a booster dose at 15 months. This setting allows the evaluation of IPV immunogenicity in a scenario where the circulation of any poliovirus is highly unlikely.

Infants will receive two or three doses of full dose IPV IM or fractional dose f-IPV ID, in various schedule combinations (6 and 14 weeks; 10 and 14 weeks; 14 and 36 weeks; 6, 14 and 36 weeks; 10, 14 and 36 weeks). Immunological and safety assessments will be made after one dose, two doses and three doses.

The study will be conducted in Montevideo, Uruguay and a total of 1493 infants will be randomized into 6 groups. Other vaccines comprise DTPw-HB-Hib (pentavalent combined diphtheria-tetanus-whole cell pertussis-hepatitis B-Hib vaccine), Pneumococcal conjugate vaccine, Rotavirus and will be administered concomitantly.

Optimum immunogenicity expected from the dose/s of IPV in the post-eradication era will have to be balanced with the cost and supply constraints of IPV. This study will be critical to determine how many doses of IPV and which schedule will be recommended for the post-eradication era after the cessation of OPV (oral polio vaccine) usage globally.

ELIGIBILITY:
Inclusion Criteria:

* Infants of 6 weeks of age (-7 to + 7 days) on date of first vaccination
* Healthy, as assessed from medical history and physical examination by a study physician
* Written informed consent obtained from parents or legal representatives that they have been properly informed about the study and are able to comply with planned study procedures

Exclusion Criteria:

* Vaccinated with any poliovirus vaccine prior to inclusion
* A household contact with OPV vaccination history in the past 4 weeks
* HIV infection or pharmacologic immunosuppression.
* Known allergy to any component of the study vaccines (phenoxyethanol, formaldehyde)
* Uncontrolled coagulopathy or blood disorder contraindicating intramuscular and intradermal injections.
* Acute severe febrile illness on day of vaccination deemed by the Investigator to be a contraindication for vaccination.
* Not suitable for inclusion or is unlikely to comply with the protocol in the opinion of the investigator.

Ages: 5 Weeks to 7 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Seroconversion | To be assessed four weeks after the second vaccination for all groups receiving 2 doses of IPV and four weeks after the second vaccination for all groups receiving 2 doses of f-IPV.
  Seroconversion will be defined as a change from seronegative to seropositive (antibody titers of ≥1:8) and in infants seropositive at baseline (assumed to be from maternally-derived antibody titers), as a ≥4-fold rise in antibody titers post-vaccination, computed by assuming an exponential decay model with a half-life of 24 days.

SECONDARY OUTCOMES:
Seroconversion | To be assessed four weeks after the second or third vaccination, respectively, for the groups receiving IPV and four weeks after the second or third vaccination, respectively, for the groups receiving f-IPV.
Median titers | To be assessed four weeks after the second or third vaccination, respectively, for the groups receiving IPV and four weeks after the second or third vaccination, respectively, for the groups receiving f-IPV.
SAEs (Serious Adverse Events) | To be assessed throughout the complete study period, approx. 18 months.
IMEs (Important Medical Events) | To be assessed throughout the complete study period, approx. 18 months.
  These are medically significant events that do not meet any of the SAE criteria, but require medical or surgical consultation or intervention to prevent this event from becoming a SAE.
Severe local reactions | To be assessed throughout the complete study period, approx. 18 months.
  Severe local reactions can include severe pain, inflammation, induration and edema in the injection area.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Gutierrez, MD, Principal Investigator — CASMU Polyclinic 8 de Octubre 3310 Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: Undecided